CLINICAL TRIAL: NCT00654680
Title: A Rand, db, Parallel-group, Plac-controlled Study Evaluating the Efficacy and Safety of Vardenafil Administered for 12 Weeks in a Flexible-dose Regimen Compared to Plac in Subjects With ED Solely Secondary to Traumatic Spinal Cord Injury
Brief Title: Evaluating the Efficacy and Safety of Vardenafil in Patients Erectile Dysfunction Solely Secondary to Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10473
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Traumatic spinal cord injury; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Vardenafil (Levitra, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil (Levitra, BAY38-9456) — 5mg, 10mg or 20mg taken 1 hour prior to sexual intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
Investigate efficacy and safety of Vardenafil in patients with spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* Males ≥18 years with erectile dysfunction (ED) solely as a result of traumatic spinal cord injury (SCI) for ≥6 months with demonstrated 50% failure in intercourse attempts during the 4-week run-in period.
* Stable heterosexual relationship for at least 1 month.

Exclusion Criteria:

* Subjects with unstable medical or psychiatric conditions or using prohibited concomitant medications
* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy
* Other exclusion criteria apply according to US Product Information or Summary of Product Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2002-10; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function-Erectile Function domain | 12 weeks

SECONDARY OUTCOMES:
Sexual Encounter Profile Question 2 | 12 weeks
Sexual Encounter Profile Question 3 | 12 weeks
Other diary based variables | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer